CLINICAL TRIAL: NCT07003828
Title: Hemodialysis-Induced Renal Perfusion Decline: Unraveling the Pathophysiological Mechanisms Linking Intradialytic Circulatory Stress to Residual Renal Function Loss
Acronym: HD-RPD
Status: Active, not recruiting | Type: Observational
Sponsor: Yuanjun Yang (Other)
Responsible Party: Sponsor-Investigator, Yuanjun Yang, doctor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: S2024-294-01
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: End-Stage Renal Disease Requiring Haemodialysis
Keywords: hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients with end-stage renal disease (ESRD) within 3 months of commencing HD
  Interventions: Diagnostic Test: CEUS examinations

INTERVENTIONS:
Diagnostic Test: CEUS examinations — CEUS examinations were performed at three predetermined time points during each HD session: immediately before, 3 hours after HD initiation, and 15 minutes post-dialysis.

SUMMARY:
Residual renal function (RRF) plays a critical role in quality of life and survival in hemodialysis (HD) patients but characteristically declines after the initiation of HD. Owing to incomplete understanding of the pathophysiology underlying RRF decline, protective strategies remain limited. The aim of this study was to characterize the changes in renal perfusion in incident HD patients with preserved RRF during dialysis sessions and to provide new strategies for RRF preservation.

ELIGIBILITY:
Inclusion Criteria:

* (1) adult patients with end-stage renal disease (ESRD) within 3 months of commencing HD; (2) preserved RRF defined as urinary output >500 mL/24 h or eGFR ≥3 mL/min/1.73 m²

Exclusion Criteria:

* (1) known allergy to sulfur hexafluoride microbubbles (SonoVue®) microbubbles; (2) vascular access dysfunction; (3) combined peritoneal dialysis; (4)severe cardiopulmonary disease; (5) active infection or malignancy; (6) communicable diseases; (7) pregnancy or breastfeeding; (8) participation in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of thirty patients from the First Medical Center of Chinese PLA General Hospital were consecutively enrolled in the study (as detailed in the Study Design section) after providing written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Renal perfusion | at three time points during the HD session: pre-dialysis baseline, intradialytic phase (3 hours post-initiation)
  Renal perfusion was quantified using the CEUS-assessed perfusion index (PI). The primary outcome measure was the PI.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Medical Center of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie D, Tan J, Zhang Q, Yu Q, Wang Y, Wang Y, Gao L, Yan L, Zhou J, Li N, Cai G. Hemodialysis-induced renal perfusion decline: unraveling the pathophysiological mechanisms linking intradialytic circulatory stress to residual renal function loss. Front Pharmacol. 2025 Oct 20;16:1648608. doi: 10.3389/fphar.2025.1648608. eCollection 2025. PMID 41190031